CLINICAL TRIAL: NCT06998758
Title: Megestrol Acetate in Improving Neoadjuvant Chemotherapy-Related Weight Loss in Patients With Locally Advanced Colorectal Cancer: A Multicenter Randomized Controlled Clinical Trial
Brief Title: Megestrol Acetate in Improving Neoadjuvant Chemotherapy-Related Weight Loss in Locally Advanced CRC
Acronym: MATRIX
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jun Huang, Professor, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2025078
Record Dates: First submitted 2025-05-08; First posted 2025-05-31 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Neoadjuvant Chemotherapy; Weight Loss
Keywords: Megestrol Acetate
MeSH Terms: conditions — Weight Loss | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6 + Megestrol Acetate (Experimental): Patients from experimental group receive six cycles of neoadjuvant chemotherapy with mFOLFOX6 (oxaliplatin 85 mg/m², leucovorin calcium 400 mg/m², fluorouracil 400 mg/m², and fluorouracil 2400 mg/m² continuous infusion over 48 hours on day 1) every 2 weeks and megestrol acetate at 625 mg/day by oral until the end of neoadjuvant chemotherapy.
  Interventions: Drug: Megestrol Acetate
- mFOLFOX6 (No Intervention): Patients from this group receive six cycles of neoadjuvant chemotherapy with mFOLFOX6 (oxaliplatin 85 mg/m², leucovorin calcium 400 mg/m², fluorouracil 400 mg/m², and fluorouracil 2400 mg/m² continuous infusion over 48 hours on day 1) every 2 weeks

INTERVENTIONS:
Drug: Megestrol Acetate — Oral megestrol acetate at 625 mg/day is given from the beginning to the end of neoadjuvant chemotherapy.
  Arms: mFOLFOX6 + Megestrol Acetate

SUMMARY:
Cancer-associated anorexia, a debilitating condition characterized by progressive appetite loss in oncology patients, contributes to pancytopenia, sarcopenia, and adipose tissue depletion. Megestrol acetate (MA) improves appetite and promotes weight gain through multiple mechanisms, playing a crucial role in the nutritional management of cancer patients. Total mesorectal excision (TME) following neoadjuvant chemotherapy has become the standard treatment strategy for patients with locally advanced colorectal cancer (LACRC). Despite its oncological benefits, neoadjuvant chemotherapy frequently induces grade ≥2 gastrointestinal toxicities (including nausea, emesis, and diarrhea) that exacerbate malnutrition through appetite suppression and negative energy balance. Previous studies have demonstrated that combining MA with first-line maintenance chemotherapy in patients with metastatic colorectal cancer significantly improves appetite, increases body weight, enhances quality of life, and improves prognosis. However, the safety and efficacy of MA during the neoadjuvant treatment phase of LACRC remain unclear. This multicenter, randomized controlled clinical trial aims to evaluate the effects of MA on chemotherapy--related weight loss, anorexia, nutritional status, and chemotherapy tolerance in patients with LACRC undergoing neoadjuvant chemotherapy. Additionally, this study will assess the safety profile of MA in this clinical setting.

DETAILED DESCRIPTION:
This clinical trial is an open-label, prospective, multicenter, randomized study. The aims of this study are to evaluate the effects of megestrol acetate (MA) on ameliorating neoadjuvant chemotherapy-related weight loss, anorexia, nutritional deterioration, andChemotherapy-related adverse events in patients with locally advanced colorectal cancer (LACRC), while comprehensively assessing its safety profile. Eligible participants will be randomly assigned in a 1:1 ratio to either the experimental group or the control group. Participants in the experimental group will receive 6 cycles of neoadjuvant chemotherapy regimen of mFOLFOX6 (intravenous oxaliplatin 85 mg/m2, leucovorin 400 mg/m2, 5-fluorouracil 400 mg/m2, and 5-fluorouracil 2400 mg/m2 continuous pumping for 48 hours) administered every 14 days, combined with oral MA suspension at a dose of 625 mg/day. MA treatment will be maintained until the completion of neoadjuvant chemotherapy. Participants in the control group will receive 6 cycles of the mFOLFOX6 neoadjuvant chemotherapy regimen without concurrent administration of MA. Subjects in both the experimental and control groups will undergo radical surgical treatment after completing the neoadjuvant therapy. Those achieving pCR based on postoperative pathology will be regularly followed up according to the follow-up protocol. Participants who do not achieve pCR will receive six cycles of adjuvant therapy after surgery, followed by regular follow-up assessments as outlined in the protocol after completing the final cycle of adjuvant therapy. The primary outcome of this study is the incidence of weight loss (defined as >5% body weight reduction during neoadjuvant therapy). Secondary objectives include: 1) Appetite evaluation; 2) Nutritional parameter dynamics; 3) Quality of life (QoL) assessment with the EORTC QLQ-C30 questionnaire; 4) Incidence of neoadjuvant chemotherapy-related adverse events; 5) Oncological response; 6) Surgical morbidity; 7) Postoperative recovery metrics: time to first flatus/bowel movement, length of postoperative hospitalization, and 30-day readmission rates; 8) Survival outcomes: 1-year disease-free survival (DFS), Overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females aged between 18 and 75 years old.
* Histologically confirmed colorectal adenocarcinoma.
* Immunohistochemistry showing pMMR or MSI status determined as MSS.
* Clinical stage cTxN1-2M0, with or without MRF positivity, and with or without EMVI positivity.
* ECOG performance status 0-1, with a life expectancy of ≥6 months.
* Deemed suitable for preoperative mFOLFOX6 neoadjuvant chemotherapy following multidisciplinary team discussion.
* Written informed consent has been obtained from the patients.

Exclusion Criteria:

* Patients with cardiac arrhythmias requiring anti-arrhythmic treatment (excluding β-blockers or digoxin), symptomatic coronary artery disease or myocardial ischemia (myocardial infarction within the past 6 months), or congestive heart failure greater than NYHA Class II.
* Patients with poorly controlled severe hypertension.
* Patients with a history of HIV infection or active chronic hepatitis B or C (with high-copy viral DNA).
* Patients with active tuberculosis (TB) who are receiving anti-tuberculosis treatment or have received anti-tuberculosis treatment within 1 year prior to screening.
* Patients with other active severe clinical infections (per NCI-CTC v.5.0).
* Patients who have previously received chemotherapy.
* Patients with a history of seizures requiring treatment (e.g., steroids or anti-epileptic therapy).
* Patients with drug abuse or medical, psychological, or social conditions that may interfere with study participation or outcome assessment.
* Patients with a known or suspected allergy to the study drug or any agents administered in relation to the trial.
* Patients with any unstable condition that may jeopardize patient safety or compliance.
* Pregnant or breastfeeding women, or fertile women not using adequate contraception.
* Patients who refuse to sign the informed consent form.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2027-05-10 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of weight loss | 1 year
  the rate of weight loss

SECONDARY OUTCOMES:
Appetite assessment | 1 year
  Questionnaire to assess appetite of patients based on the FAACT-A/CS(Functional Assessment of Anorexia/ Cachexia Therapy) scale. A total score of more than 37 indicates a good appetite. A total score of 37 or less suggests loss of appetite, with lower scores indicating more severe anorexia.
Changes in nutritional indicators | 1 year
  Nutritional indicators including serum albumin and pre-albumin
Quality of life assessment | 1 year
  questionnaire to assess quality of life based on the EORTC(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire) QLQ-C30 scale，ranged from 0 to 100. The higher the patient's score, the better their quality of life.
AEs related to NCT | 1 year
  Incidence of adverse events related to neoadjuvant chemotherapy
Tumor response assessment of neoadjuvant chemotherapy | 1 year
  Standardized framework for evaluating the efficacy of cancer treatments by RECIST 1.1
AEs related to surgery | 1 year
  Incidence of adverse events related to surgery
Time to first flatus | 1 year
  Time to first flatus after surgery, indicator of postoperative recovery
Time to first defecation | 1 year
  Time to first defecation after surgery, indicator of postoperative recovery
Postoperative hospital stays | 1 year
  Duration in hospital after surgery, indicator of postoperative recovery
1 year of DFS | 1 year
  1-year disease-free survival
1 year OS | 1 year
  1-year overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Jun Huang, PhD., Principal Investigator — Sun Yat-sen University
Locations (1):
- The Sixth Affiliated Hospital of Sun-Yat sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided